CLINICAL TRIAL: NCT02760680
Title: Validierung Der Peripher Arteriellen Tonometrie Zur Diagnostik Schlafbezogener Atmungsstörungen Bei Patienten Mit Systolischer Herzinsuffizienz
Brief Title: Validation of the Peripheral Arterial Tone to Detect Sleep-disordered Breathing in Patients With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Collaborators: Itamar-Medical, Israel (Industry)
Responsible Party: Principal Investigator, Thomas Bitter, Dr. med, Heart and Diabetes Center North-Rhine Westfalia
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: HDZNRW-KA_005_TB
Record Dates: First submitted 2016-04-20; First posted 2016-05-04 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Sleep-Disordered Breathing
Keywords: Chronic Heart Failure; Sleep-Disordered Breathing; Peripheral Arterial Tone
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polysomnography (Placebo Comparator): The PSG is known as the "Gold Standard" for detecting SDB: experienced sleep physicians and technicians score events (apnea/hypopnea) using current AASM Guidelines.
  Interventions: Device: WatchPAT 200 (TM); Other: Polysomnography
- Diagnostic Device (WatchPAT 200 (TM)) (Active Comparator): The WatchPAT 200 (TM) is a wrist worn diagnostic device for detecting SDB. Its main part is the measurement of the peripheral arterial tone (PAT) via a plethysmographic based finger-mounted probe. It can measure the level of sympathetic activation of the autonomic nervous system. Pulse rate, oxygen saturation and snoring/body position levels are calculated, too. A software program (zzzPAT (TM)) with a special algorithm analyzes the raw data and creates a sleep report. Therefore the property of the WatchPAT 200 (TM) proclaims that the WatchPAT 200 (TM) can detect sleep events and SDB.
  Interventions: Device: WatchPAT 200 (TM); Other: Polysomnography

INTERVENTIONS:
Device: WatchPAT 200 (TM) — The WatchPAT 200 (TM) is a wrist worn diagnostic device for detecting SDB. Its main part is the measurement of the peripheral arterial tone (PAT) via a plethysmographic based finger-mounted probe. It can measure the level of sympathetic activation of the autonomic nervous system. Pulse rate, oxygen saturation and snoring/body position levels are calculated, too. A software program (zzzPAT (TM)) with a special algorithm analyzes the raw data and creates a sleep report. Therefore the property of the WatchPAT 200 (TM) proclaims that the WatchPAT 200 (TM) can detect sleep events and SDB.
  Other Names: PAT (TM) - Watch-PAT 200, Itamar-Medical Ltd., Israel
Other: Polysomnography — The PSG is known as the "Gold Standard" for detecting SDB: experienced sleep physicians and technicians score events (apnea/hypopnea) using current AASM Guidelines.

SUMMARY:
A prospective validation study: Level I-full night-polysomnography (PSG) versus a diagnostic device with measurement of the peripheral arterial tone (PAT) of patients with chronic heart failure (CHF) and sleep-disordered breathing (SDB).

DETAILED DESCRIPTION:
Patients with chronic heart failure (CHF), reduced left ventricular ejection fraction (LVEF<45%) and predicted sleep-disordered breathing (SDB) receive a diagnostic device (WatchPAT 200 (TM)) and polysomnography (PSG) simultaneously during on night in a hospital sleep lab.

The WatchPAT 200 (TM) is a wrist worn diagnostic device for detecting SDB. Its main part is the measurement of the peripheral arterial tone (PAT) via a plethysmographic based finger-mounted probe. It can measure the level of sympathetic activation of the autonomic nervous system. Pulse rate, oxygen saturation and snoring/body position levels are calculated, too. A software program (zzzPAT (TM)) with a special algorithm analyzes the raw data and creates a sleep report. Therefore the property of the WatchPAT 200 (TM) proclaims that the WatchPAT 200 (TM) can detect sleep events and SDB.

The PSG is scored by sleep lab physicians/technicians blinded to the zzzPAT (TM)-software results using current American Academy of Sleep Medicine (AASM) guidelines.

Both results will be compared and the results of the device will be validated and evaluated against the results of the "Gold Standard" polysomnography.

ELIGIBILITY:
Inclusion Criteria:

* reduced left ventricular ejection fraction (LVEF) < 45 %
* indication for a polysomnography

Exclusion Criteria:

* allergies against the device or parts of the device
* psychogenic or neurological disorders which do not allow a sufficient patient compliance
* osteogenetic disorders which do not allow a painless investigation
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Apnea-Hypopnea-Index (AHI) | one night of sleep
  Index is stated per hour (/h)

SECONDARY OUTCOMES:
Sleep: Time in bed | one night of sleep
  stated in minutes (min)
Sleep: Total sleep time | one night of sleep
  stated in minutes (min)
Sleep: Sleep latency | one night of sleep
  stated in minutes (min)
Sleep: Rapid-Eye-Movement (REM) sleep latency | one night of sleep
  stated in minutes (min)
Sleep: latency to S3 | one night of sleep
  stated in minutes (min)
Sleep: Wake | one night of sleep
  stated in percent (%)
Sleep: S1 stadium/total sleep time | one night of sleep
  stated in percent (%)
Sleep: S2 stadium/total sleep time | one night of sleep
  stated in percent (%)
Sleep: S3 stadium/total sleep time | one night of sleep
  stated in percent (%)
Sleep: REM sleep/total sleep time | one night of sleep
  stated in percent (%)
Sleep: Sleep Efficiency | one night of sleep
  amount of sleep, stated in percent (%)
Sleep: Number of Wakes | one night of sleep
  stated as number
Respiratory Parameters: Oxygen-Desaturation-Index (ODI) | one night of sleep
  Index is stated per hour (/h)
Respiratory Parameters: longest Apnea | one night of sleep
  stated in seconds (s)
Respiratory Parameters: longest Hypopnea | one night of sleep
  stated in seconds (s)
Respiratory Parameters: Obstructive Apnea | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Central Apnea | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Mixed Apnea | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Obstructive Hypopnea | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Central Hypopnea | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Hypopnea total | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Apnea + Hypopnea total | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Desaturations | one night of sleep
  Index is stated per hour (/h), stated as number
Respiratory Parameters: Mean Oxygen Saturation (sO2) | one night of sleep
  stated in percent (%)
Respiratory Parameters: Minimum Oxygen Saturation (sO2) | one night of sleep
  stated in percent (%)
Respiratory Parameters: Maximum Oxygen Saturation (sO2) | one night of sleep
  stated in percent (%)
Respiratory Parameters: Mean of Desaturations Nadirs | one night of sleep
  stated in percent (%)
Respiratory Parameters: Mean of Desaturations | one night of sleep
  stated in percent (%)
Respiratory Parameters: Time Oxygen Saturation (TsO2) < 90% | one night of sleep
  stated in percent (%), stated in minutes (min)
Respiratory Parameters: Respiratory-Disturbance-Index (RDI) | one night of sleep
  Index is stated per hour (/h)
Differences of results of patients with central sleep apnea (CSA) or obstructive sleep apnea (OSA) | one night of sleep
  Comparison of all Parameters added above

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bitter, MD, Study Director — Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany; Florian Schindhelm, Principal Investigator — Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany
Locations (1):
- Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Bad Oeynhausen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bar A, Pillar G, Dvir I, Sheffy J, Schnall RP, Lavie P. Evaluation of a portable device based on peripheral arterial tone for unattended home sleep studies. Chest. 2003 Mar;123(3):695-703. doi: 10.1378/chest.123.3.695. PMID 12628865
- See also: Official website of Herz- und Diabeteszentrum NRW, Ruhr-Universitaet Bochum, Bad Oeynhausen, Germany — http://www.hdz-nrw.de
- See also: Official website of Itamar Medical Ltd. — http://www.itamar-medical.com